CLINICAL TRIAL: NCT02343588
Title: Development and Application of Appropriate Technology for Obesity Prevention and Control in Seven Centers in China
Brief Title: A National School-based Health Lifestyles Interventions Among Chinese Children and Adolescents Against Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Peking University (Other); Central South University (Other); Tianjin Medical University (Other); Shanghai Municipal Center for Disease Control and Prevention (Other); Chongqing Medical University (Other); Ningxia Medical University (Other)
Responsible Party: Principal Investigator, CHEN Yajun, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201202010
Record Dates: First submitted 2015-01-07; First posted 2015-01-22 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Pediatric Obesity
Keywords: Chinese multi-centered school based obesity intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Health Lifestyles Interventions (Experimental): 1. Creating a supportive school, family and community environment;
  2. Health lifestyles educational strategies;
  3. Instruct and promote school physical education;
  4. The monitoring and instruction of obesity related behaviors (focus group)
  Interventions: Behavioral: The Health Lifestyles Interventions
- Receive no intervention (No Intervention): Usual practice

INTERVENTIONS:
Behavioral: The Health Lifestyles Interventions — 1. Creating supportive school and family environment, whole intervention periods;
  2. Health lifestyles educational strategies, 30min/week for education lessons and six times education activities;
  3. Instruct and promote school physical education, whole intervention periods;
  4. The monitoring and instruction of obesity related behaviors, once a week for physical activity and dietary behavioral log and once a month for parental monitor
  Arms: The Health Lifestyles Interventions

SUMMARY:
The study was designed as a national multi-centered cluster randomized controlled trial involving more than 70,000 children and adolescents aged 7-18 years from 7 provinces in China. In each center, about 12-16 primary and secondary schools, with totally at least 10000 participants were randomly selected (Primary: Secondary=1:1). All of the selected schools were randomly allocated to either intervention or control group (Intervention: Control=1:1).The multi-components school-based and family-involved scheme was conducted within the intervention group for 9 month, while students in the control group followed their usual health practice. The intervention consisted of four components: a) Create supportive school and family environment, b) Health lifestyles education and related compulsory physical activities, c) Instruct and promote school physical education, d) Self-monitor obesity related behaviors. Four types of outcomes including anthropometric, behavioral, blood chemical and physical fitness were measured to assess the effectiveness of the intervention program.

ELIGIBILITY:
Inclusion Criteria:

grade of 1 to 5 in primary schools and grade of 6 to 8 and 10 to 11 in secondary schools.

Exclusion Criteria:

Suffering or any history of disabilities, cardiovascular diseases, asthma, metabolic diseases, etc.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70000 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in the prevalence of overweight and obesity | Baseline, Month 9

SECONDARY OUTCOMES:
Change in obesity related anthropometric measurements (waist circumference, hip circumference, blood pressure and skin fold thickness) | Baseline, Month 9
Change in physical activity and dietary behaviors (Dietary, sedentary or physical activity behaviors and their determents, as measured by validated questionnaires (parent, children and school version) | Baseline, Month 9
Change in serum lipids and fasting glucose (fasting plasma glucose, fasting triglycerides, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol) | Baseline, Month 9
Change in physical fitness (standing-board jump, 50 meters speed run, 50 meters × 8 shuttle run (primary students) and run 800/1000 meters (secondary school students) | Baseline, Month 9

CONTACTS AND LOCATIONS:
Overall Officials: Jun MA, M.D, Study Chair — Peking University; Jiayou LUO, M.D, Principal Investigator — Central South University; Xin ZHANG, M.D, Principal Investigator — Tianjin Medical University; Chunyan LUO, M.D, Principal Investigator — Shanghai Municipal Center for Disease Control and Prevention & Shanghai Institutes of Preventive Medicine; Hong WANG, M.D, Principal Investigator — Chongqing Medical University; Haiping ZHAO, M.D, Principal Investigator — Ningxia Medical University; Dehong PAN, M.D, Principal Investigator — Liaoning Health Supervision Bureau; Jin JING, M.D, Principal Investigator — Sun Yat-sen University

REFERENCES:
- [Derived] Guo P, Zhou Y, Zou Z, Chen Y, Jing J, Ma Y, Song Y, Ling W, Ma J, Zhu Y. Effects of School-Based Lifestyle Interventions on Cardiovascular Health in Chinese Children and Adolescents: A Post Hoc Analysis of a National Multicenter Study. J Am Heart Assoc. 2025 Jan 7;14(1):e037371. doi: 10.1161/JAHA.124.037371. Epub 2024 Dec 20. PMID 39704211
- [Derived] Guo P, Zhou Y, Zhu Y. Effects of a school-based lifestyle intervention on ideal cardiovascular health in Chinese children and adolescents: a national, multicentre, cluster-randomised controlled trial. Lancet Glob Health. 2023 Mar;11 Suppl 1:S14. doi: 10.1016/S2214-109X(23)00097-9. PMID 36866471
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Dong Y, Zou Z, Wang H, Dong B, Hu P, Ma Y, Song Y, Ma J. National School-Based Health Lifestyles Intervention in Chinese Children and Adolescents on Obesity and Hypertension. Front Pediatr. 2021 May 28;9:615283. doi: 10.3389/fped.2021.615283. eCollection 2021. PMID 34123956
- [Derived] Diao H, Wang H, Yang L, Li T. The impacts of multiple obesity-related interventions on quality of life in children and adolescents: a randomized controlled trial. Health Qual Life Outcomes. 2020 Jul 6;18(1):213. doi: 10.1186/s12955-020-01459-0. PMID 32631401
- [Derived] Zou Z, Yang Z, Yang Z, Wang X, Gao D, Dong Y, Ma J, Ma Y. Association of high birth weight with overweight and obesity in Chinese students aged 6-18 years: a national, cross-sectional study in China. BMJ Open. 2019 May 22;9(5):e024532. doi: 10.1136/bmjopen-2018-024532. PMID 31122966